CLINICAL TRIAL: NCT04284202
Title: PD-1 Combined With Dasatinib for as Third-line Treatment for ARID1A Mutation Advanced NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, zhangxiaochun, Director of Precision Medicine Center, The Affiliated Hospital of Qingdao University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOT-ARID1A
Record Dates: First submitted 2020-02-23; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: NSCLC Stage IV; ARID1A; PD-1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PD-1 plus Dasatinib (Experimental)
  Interventions: Drug: PD-1 plus Dasatinib

INTERVENTIONS:
Drug: PD-1 plus Dasatinib — Toripalimub 240mg injection day1; Dasatinib 100mg po qd day1-day21. 3weeks is 1 cycle.

SUMMARY:
The purpose of this study is to evalute the efficacy and safety of PD-1 antibody combined with Dasatinib as third-line therapy for NSCLC patients with ARID1A mutation until disease progression or intolerable toxicity or patients withdrawal of consent. The target sample size is 30+individuals. The primary endpoint of this study is PFS、ORR、OS and the secondary endpoint is toxicity.

ELIGIBILITY:
Inclusion Criteria:

- 1. Provision of signed and dated written informed consent by the patient or legally acceptable representative prior to any study-specific procedures 2. over 18 years old 3. Metastatic (stage IV) NSCLCwith ARID1A mutation underwent 2 lines of prior treatment.

4. World Health Organization (WHO) performance status 0-2 5. Adequate bone marrow reserve and organ function as demonstrated by complete blood count, biochemistry in blood and urine at baseline 6. ECG recording at baseline showing absence of any cardiac abnormality as per exclusion criterion #5 7. Female patients of childbearing potential must be using adequate contraceptive measures must not be breast feeding, and must have a negative pregnancy test prior to start of dosing.

Exclusion Criteria:

- 1. Subjects with known EGFR and ALK mutations are excluded. 2. Subjects with untreated CNS metastases are excluded 3. Subjects with an active, known or suspected autoimmune disease. 4. Prior therapy with an anti-PD-1, anti-PD-L1, anti-PDL-2, or anti-CTLA-4 antibody or any other antibody targeting T cell co-regulatory pathways.

5. Prior therapy with Dasatinib 6. Known medical condition that, in the investigator's opinion, would increase the risk associated with study participation or study drug administration or interfere with the interpretation of safety results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Event driven, an expected average of 6 months

SECONDARY OUTCOMES:
Overall survival(OS) | An expected average of 24months

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, China

IPD SHARING:
Plan to Share IPD: No